CLINICAL TRIAL: NCT06827613
Title: A Phase 1b/2, Open-label Study to Investigate the Safety and Efficacy of Invikafusp Alfa (STAR0602), a Selective T Cell Receptor (TCR)-Targeting, Bifunctional Antibody-fusion Molecule, in Combination With Sacituzumab Govitecan in Participants With Unresectable, Locally Advanced, or Metastatic Solid Tumors (START-002)
Brief Title: A Study of Invikafusp Alfa (STAR0602), a Selective T Cell Receptor (TCR)-Targeting, Bifunctional Antibody-fusion Molecule, in Combination With Sacituzumab Govitecan in Participants With Advanced Solid Tumors
Acronym: START-002
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Marengo Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: START-002
Record Dates: First submitted 2025-01-28; First posted 2025-02-14 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Triple Negative Locally Advanced Non-resectable Breast Cancer; HR+, HER2-, Advanced Breast Cancer
MeSH Terms: interventions — sacituzumab govitecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase 1 Safety Run-In: Advanced Solid Tumors (Experimental): Interventions: STAR0602 + Sacituzumab Govitecan
  Interventions: Drug: STAR0602; Drug: Sacituzumab Govitecan (SG)
- Phase 2 Cohort Expansion: Advanced Solid Tumors (Experimental): Interventions: STAR0602 + Sacituzumab Govitecan at the Recommended Expansion Dose (RED) from Phase 1
  Interventions: Drug: STAR0602; Drug: Sacituzumab Govitecan (SG)

INTERVENTIONS:
Drug: STAR0602 — solution, intravenous infusion
Drug: Sacituzumab Govitecan (SG) — intravenous infusion, 10mg/kg

SUMMARY:
This is a Phase 1b/2, Open-label Study to Investigate the Safety and Efficacy of Invikafusp alfa (STAR0602), a Selective T Cell Receptor (TCR)-targeting, Bifunctional Antibody-fusion Molecule, in Combination with Sacituzumab Govitecan in Participants with Unresectable, Locally Advanced, or Metastatic Solid Tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Have measurable disease as per RECIST v1.1 criteria and documented by CT and/or MRI. Cutaneous or subcutaneous lesions must be measurable by calipers.
2. Tumor Type:

   * mTNBC (Safety Run-in and Cohort A): Progression or recurrence of locally advanced or metastatic TNBC
   * HR+/HER2- mBC (Safety Run-in and Cohort B): Progression or recurrence of locally advanced or metastatic HR+/HER2- breast cancer
3. Symptomatic central nervous system (CNS) metastases must have been treated, be asymptomatic for ≥ 14 days, and meet the following at the time of enrollment:

No concurrent treatment for CNS disease (eg, surgery, radiation, corticosteroids > 10 mg prednisone/day or equivalent); No concurrent leptomeningeal disease or cord compression.

Exclusion Criteria:

1. History of known autoimmune disease with exceptions of:

   * Vitiligo
   * Psoriasis
   * Atopic dermatitis or other autoimmune skin condition not requiring systemic treatment
   * History of Graves' disease, now euthyroid for > 4 weeks
   * Hypothyroidism managed by thyroid replacement
   * Alopecia
   * Arthritis managed without systemic therapy beyond oral nonsteroidal anti-inflammatory drugs
   * Adrenal insufficiency well-controlled on replacement therapy
2. Major surgery or traumatic injury within 8 weeks before first dose of study intervention
3. Unhealed wounds from surgery or injury
4. Clinically significant cardiovascular/vascular disease, gastrointestinal disorders, inflammatory processes, pulmonary compromises
5. Active viral, bacterial, or systemic fungal infection requiring parenteral treatment within 7 days prior to the initiation of study intervention.
6. Vaccination with any live virus vaccine within 4 weeks prior to the initiation of study intervention administration. Inactivated annual influenza vaccination is allowed.
7. Participants who are known to be human immunodeficiency virus positive or hepatitis B or C positive and have uncontrolled disease.
8. Second primary invasive malignancy not in remission for ≥ 1 year. Exceptions include non-melanoma locally advanced skin cancer, cervical carcinoma in situ, localized prostate cancer (Gleason score ≤ 7), resected melanoma in situ, or any malignancy considered to be indolent and never required systemic therapy, with the exception of indolent lymphomas.
9. Pregnant, likely to become pregnant, or lactating women (where pregnancy is defined as the state of a female after conception and until the termination of gestation)
10. Treatment with >10 mg per day of prednisone (or equivalent) or other immune-suppressive drugs within 7 days prior to the initiation of study intervention. Exceptions may be made for participants who have had allergic reactions to iodinated contrast media. Steroids for topical, ophthalmic, inhaled, or nasal administration are allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-03-24 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Phase 1 (Safety Run-In): Number of Participants with Dose Limiting Toxicites (DLTs) | 21 days following the first dose of STAR0602 + Sacituzumab Govitecan
Phase 1 and 2 (Safety Run-In and Cohort Expansion): Number of Participants with Adverse Events and Serious Adverse Events | Up to 3 years
Phase 1 and 2 (Safety Run-In and Cohort Expansion): Percentage of participants with Overall Objective Tumor Responses (ORR) | Up to 3 years
  Proportion of participants who have a complete response (CR) or partial response (PR)

SECONDARY OUTCOMES:
Phase 1 and 2 (Safety Run-In and Cohort Expansion): Duration of Response (DOR) | Up to 3 years
Phase 1 and 2 (Safety Run-In and Cohort Expansion): Percentage of Participants with Disease Contral (DCR) | Up to 3 years
  Proportion of participants who have a complete response (CR) or partial response (PR) or stable disease (SD)
Phase 1 and 2 (Safety Run-In and Cohort Expansion): Progression Free Survival (PFS) | Up to 3 years
Phase 1 and 2 (Safety Run-In and Cohort Expansion): Overall Survival (OS) | Up to 3 years
Phase 1 and 2 (Safety Run-In and Cohort Expansion): Maximum Observed Concentration (Cmax) for STAR0602 | Cycle 1 and Cycle 3 at predefined intervals (Cycle length = 21 days) up to 3 years
Phase 1 and 2 (Safety Run-In and Cohort Expansion): Area Under the Concentration Curve (AUC) for STAR0602 | Cycle 1 and Cycle 3 at predefined intervals (Cycle length = 21 days) up to 3 years
Phase 1 and 2 (Safety Run-In and Cohort Expansion): Apparent Total Body Clearance (CL) for STAR0602 | Cycle 1 and Cycle 3 at predefined intervals (Cycle length = 21 days) up to 3 years
Phase 1 and 2 (Safety Run-In and Cohort Expansion): Apparent Volume of Distribution (Vd) for STAR0602 | Cycle 1 and Cycle 3 at predefined intervals (Cycle length = 21 days) up to 3 years

CONTACTS AND LOCATIONS:
Locations (8):
- United States (6):
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - UCLA Health, Los Angeles, California
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - UT Health San Antonio MD Anderson Cancer Center, San Antonio, Texas
- Canada (2):
  - BC Cancer, Vancouver, British Columbia
  - Princess Margaret Cancer Centre, Toronto, Ontario